CLINICAL TRIAL: NCT05436860
Title: Pre- Emergency / Acceptance Departments Study, Prevention in Emergency / Acceptance Departments: the Case of Hepatic Steatosis
Brief Title: PreDEA Study, Prevention in Emergency / Acceptance Departments: the Case of Hepatic Steatosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Clara Balsano, Full professor, University of L'Aquila
Other Study IDs: 61615
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Hepatic Steatosis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- presence of hepatic hyperechogenicity on ultrasound evaluation
  Interventions: Device: liver ultrasound
- absence of hepatic hyperechogenicity on ultrasound evaluation
  Interventions: Device: liver ultrasound

INTERVENTIONS:
Device: liver ultrasound — At the time of access to the emergency room, a cohort of male and female patients aged 18 or over will be consecutively recruited with green or white color coded triage.
  patients who agree to participate in the study will undergo liver ultrasound. Patients who test negative on ultrasound evaluation for liver hyperechogenicity will be part of the control group.

SUMMARY:
Our study aims to evaluate whether the Emergency Department (PS) can support the health system to improve the prevention and management of chronic inflammatory diseases and ensure actions aimed at screening, raising awareness and informing the population.

Specifically, the determination of the prevalence of a widely diffused pathology such as fatty liver disease aims to be the precursor of future pilot studies aimed at evaluating the advantages and critical issues of the PS as a prevention tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* Patients admitted to Emergency department in white or green code

Exclusion Criteria:

* Patients under 18
* Patients admitted to Emergency department in yellow or red code

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients admitted to Emergency department ,over 18, in white or green code
Sampling Method: Probability Sample
Enrollment: 20189 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the number of steatotic patients who access the emergency room - Emergency room as a tool for early diagnosis of hepatic steatosis | 12 months
  Evaluation of the effectiveness of the Emergency Department as a screening tool for the emergence of the submerged by measuring the prevalence, on the national territory, of hepatic steatosis in patients who access the emergency room.

SECONDARY OUTCOMES:
Develop new prognostic algorithms for assessing the risk of major and minor clinical events in patients with fatty liver. | 36 months
  Improve the approval rating of the service offered by the PS to the patient who has been assigned a white or green color code for triage.To develop new prognostic algorithms for assessing the risk of major and minor clinical events in patients with fatty liver.

CONTACTS AND LOCATIONS:
Locations (1):
- Clara Balsano, L’Aquila, Italy/L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No